CLINICAL TRIAL: NCT02549820
Title: Pilot Trial of Fetoscopic Endoluminal Tracheal Occlusion (FETO) in Severe Left Congenital Diaphragmatic Hernia (CDH)
Brief Title: Fetoscopic Endoluminal Tracheal Occlusion in Severe Left Congenital Diaphragmatic Hernia
Acronym: CHOP_FETO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Holly L Hedrick, MD, Principal Investigator, Professor of Surgery, Children's Hospital of Philadelphia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-011714
Record Dates: First submitted 2015-08-18; First posted 2015-09-15 (Estimated); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Congenital Diaphragmatic Hernia; Pulmonary Hypoplasia
Keywords: Congenital Diaphragmatic Hernia; Tracheal Occlusion
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- FETO in CDH (Experimental): Fetoscopic Endoluminal Tracheal Occlusion (FETO) will be performed by placing a detachable balloon inside the fetal airway and removing the balloon after several weeks. Devices: GoldBAL2 Detachable Balloon and BALTACCIBDPE100 Delivery Catheter
  Interventions: Device: GoldBAL2 Detachable Balloon and BALTACCIBDPE100 Delivery Catheter

INTERVENTIONS:
Device: GoldBAL2 Detachable Balloon and BALTACCIBDPE100 Delivery Catheter — Fetoscopic Endoluminal Tracheal Occlusion (FETO) in CDH with GoldBAL2 Detachable Balloon and BALTACCIBDPE100 Delivery Catheter

SUMMARY:
CDH is a birth defect characterized by the development, very early in gestation, of a hole in the diaphragm, the breathing muscle that separates the chest from the abdomen. As a result, the intestines and other organs in the abdomen can move into the chest and press on the developing lungs. This prevents the lungs from growing and developing normally.

In severe cases, CDH can lead to serious disease and death at birth. For these babies, treatment before birth may allow the lungs to grow enough before birth so these children are capable of surviving and thriving.

DETAILED DESCRIPTION:
Study Summary

All patients will complete a standard prenatal evaluation at the Center for Fetal Diagnosis and Treatment (CFDT) to find out if they are candidates. The standard clinical assessments include: Medical history and Physical exam, Level II ultrasound, Fetal echocardiogram, Fetal magnetic resonance imaging (MRI), and a Psychosocial assessment.

If determined eligible, patients will be extensively counseled by the CFDT Team and those who choose to participate will provide written, informed consent for study enrollment.

Up to 25 women will be enrolled in the FETO study. The mother and her unborn baby will undergo two procedures. A balloon will be placed in the unborn baby's airway between 27+0/7 - 29+6/7 gestational age. The balloon blocks the airway and remains in place until balloon removal. The timing for balloon removal will be determined by the CFDT Management Team and can occur between 34 +0/7 - 34+6/7 gestational age.

Mothers enrolled in this study must remain near the fetal center, under close supervision, from the time of balloon placement through delivery in the Garbose Family Special Delivery Unit.

Weekly prenatal monitoring will occur after the first procedure at the CFDT and planned delivery will occur in the Garbose Family Special Delivery Unit at term.

Postnatal stabilization and subsequent surgery to repair the diaphragm will take place at CHOP.

Infants will be followed at CHOP at 6 months, 12 months, and 2 years of age and then long-term in the Pulmonary Hypoplasia Program at The Children's Hospital of Philadelphia.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women age 18 years and older, who are able to consent
2. Singleton pregnancy

   Fetal:
3. Normal Karyotype or chromosomal microarray with non-pathologic variants
4. Diagnosis of Isolated Left CDH with liver up
5. Gestation at enrollment prior to 29 weeks plus 5 days
6. SEVERE pulmonary hypoplasia with Ultrasound Observed/Expected Lung-to-Head Ratio (O/E LHR) < 25%

Exclusion Criteria:

1. Pregnant women < 18 years
2. Maternal contraindication to fetoscopic surgery or severe maternal medical condition in pregnancy
3. Technical limitations precluding fetoscopic surgery
4. Rubber latex allergy
5. Preterm labor, cervix shortened (<15 mm at enrollment or within 24 hours of FETO balloon insertion procedure) or uterine anomaly strongly predisposing to preterm labor, placenta previa
6. Psychosocial ineligibility, precluding consent
7. Fetal Diaphragmatic hernia: right-sided or bilateral, major associated anomalies, isolated left-sided with the O/E LHR ≥ 25%
8. Inability to remain at FETO site during time period of tracheal occlusion, delivery and postnatal care

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2015-07; Primary Completion 2025-05-01 (Actual); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Successful balloon placement and removal. | 7 weeks
  Successful balloon placement and removal will be counted per patient. FETO insertion will be attempted up to 3 times in a single pregnant woman/ fetus.
  The maximum duration of balloon implantation, if placed at 27 weeks 0 days and removed in the 34th week, is 7 weeks. For those balloons placed later in gestation or removed earlier electively or emergently, the duration will be shorter.

CONTACTS AND LOCATIONS:
Overall Officials: Holly L Hedrick, MD, Principal Investigator — Children's Hospital of Philadelphia and the Center for Fetal Diagnosis and Treatment
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Jani JC, Nicolaides KH, Gratacos E, Valencia CM, Done E, Martinez JM, Gucciardo L, Cruz R, Deprest JA. Severe diaphragmatic hernia treated by fetal endoscopic tracheal occlusion. Ultrasound Obstet Gynecol. 2009 Sep;34(3):304-10. doi: 10.1002/uog.6450. PMID 19658113
- [Background] Deprest J, Nicolaides K, Done' E, Lewi P, Barki G, Largen E, DeKoninck P, Sandaite I, Ville Y, Benachi A, Jani J, Amat-Roldan I, Gratacos E. Technical aspects of fetal endoscopic tracheal occlusion for congenital diaphragmatic hernia. J Pediatr Surg. 2011 Jan;46(1):22-32. doi: 10.1016/j.jpedsurg.2010.10.008. PMID 21238635
- [Background] Deprest JA, Gratacos E, Nicolaides K, Done E, Van Mieghem T, Gucciardo L, Claus F, Debeer A, Allegaert K, Reiss I, Tibboel D. Changing perspectives on the perinatal management of isolated congenital diaphragmatic hernia in Europe. Clin Perinatol. 2009 Jun;36(2):329-47, ix. doi: 10.1016/j.clp.2009.03.004. PMID 19559323
- [Background] Danzer E, Hedrick HL. Controversies in the management of severe congenital diaphragmatic hernia. Semin Fetal Neonatal Med. 2014 Dec;19(6):376-84. doi: 10.1016/j.siny.2014.10.001. Epub 2014 Nov 7. PMID 25454678
- [Background] Deprest J, Brady P, Nicolaides K, Benachi A, Berg C, Vermeesch J, Gardener G, Gratacos E. Prenatal management of the fetus with isolated congenital diaphragmatic hernia in the era of the TOTAL trial. Semin Fetal Neonatal Med. 2014 Dec;19(6):338-48. doi: 10.1016/j.siny.2014.09.006. Epub 2014 Nov 11. PMID 25447987
- See also: FETO at The Children's Hospital of Philadelphia — https://www.chop.edu/centers-programs/center-fetal-diagnosis-and-treatment/fetoscopic-endoluminal-tracheal-occlusion-feto
- See also: CHOP Center for Fetal Diagnosis and Treatment — https://www.chop.edu/centers-programs/center-fetal-diagnosis-and-treatment
- See also: CHOP Pulmonary Hypoplasia Program — https://www.chop.edu/centers-programs/pulmonary-hypoplasia-program